CLINICAL TRIAL: NCT00091819
Title: A Phase 3, Randomized, Double Blind, Multinational Trial of Intravenous Telavancin Versus Vancomycin for Treatment of Complicated Gram Positive Skin and Skin Structure Infections With a Focus on Patients With Infections Due to Methicillin-resistant Staphylococcus Aureus
Brief Title: Comparison of Telavancin and Vancomycin for Complicated Skin and Skin Structure Infections With a Focus on Methicillin-resistant Staphylococcus Aureus
Acronym: ATLAS1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cumberland Pharmaceuticals (Industry)
Responsible Party: Steven Barriere, Pharm.D., Vice President, Clinical and Medical Affairs, Theravance, Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0017
Record Dates: First submitted 2004-09-17; First posted 2004-09-21 (Estimated); Results first posted 2009-12-08 (Estimated); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Staphylococcal Skin Infection
Keywords: staph; MRSA; cSSSI
MeSH Terms: conditions — Staphylococcal Skin Infections; Staphylococcal Infections | interventions — telavancin; Vancomycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Telavancin (Experimental)
  Interventions: Drug: Telavancin
- Vancomycin (Active Comparator)
  Interventions: Drug: Vancomycin

INTERVENTIONS:
Drug: Telavancin — Telavancin 10 mg/kg/day, IV for up to 14 days.
  Other Names: VIBATIV; TD-6424
  Arms: Telavancin
Drug: Vancomycin — Vancomycin 1 Gm IV q 12 hrs for up to 14 days.
  Arms: Vancomycin

SUMMARY:
Study 0017 compares the safety and effectiveness of an investigational drug, telavancin, and an approved drug, vancomycin, for the treatment of complicated skin and skin structure infections.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a diagnosis of one of the following complicated skin and skin structure infections with Methicillin Resistant Staphylococcus aureus (MRSA) either suspected or confirmed as the major cause of the infection:

  * major abscess requiring surgical incision and drainage
  * infected burn (see exclusion criteria for important qualifications)
  * deep/extensive cellulitis
  * infected ulcer (see exclusion criteria for important qualifications)
  * wound infections
* Patients must be expected to require at least 7 days of intravenous antibiotic treatment

Exclusion Criteria:

* Received more than 24 hours of potentially effective systemic (IV, IM or PO) antibiotic therapy prior to randomization
* Burns involving > 20% of body surface area or third-degree/full-thickness in nature, diabetic foot ulcers, ischemic ulcers/wounds, necrotizing fascitis, gas gangrene, or mediastinitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 862 (Actual)
Dates: Start 2005-01; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: G. Ralph Corey, MD, Principal Investigator — Duke University
Locations (1):
- Paradise Valley Hospital, 2400 E. 4th Street, National City, California, United States

REFERENCES:
- [Result] Stryjewski ME, Graham DR, Wilson SE, O'Riordan W, Young D, Lentnek A, Ross DP, Fowler VG, Hopkins A, Friedland HD, Barriere SL, Kitt MM, Corey GR; Assessment of Telavancin in Complicated Skin and Skin-Structure Infections Study. Telavancin versus vancomycin for the treatment of complicated skin and skin-structure infections caused by gram-positive organisms. Clin Infect Dis. 2008 Jun 1;46(11):1683-93. doi: 10.1086/587896. PMID 18444791
- [Result] Wilson SE, O'Riordan W, Hopkins A, Friedland HD, Barriere SL, Kitt MM; ATLAS Investigators. Telavancin versus vancomycin for the treatment of complicated skin and skin-structure infections associated with surgical procedures. Am J Surg. 2009 Jun;197(6):791-6. doi: 10.1016/j.amjsurg.2008.05.012. Epub 2008 Dec 18. PMID 19095213
- [Derived] Stryjewski ME, Barriere SL, O'Riordan W, Dunbar LM, Hopkins A, Genter FC, Corey GR. Efficacy of telavancin in patients with specific types of complicated skin and skin structure infections. J Antimicrob Chemother. 2012 Jun;67(6):1496-502. doi: 10.1093/jac/dks081. Epub 2012 Mar 13. PMID 22416054

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment Period: 19 January 2005 to 12 June 2006
Groups:
- Telavancin: Patients with complicated Gram-positive skin and skin structure infections (primarily due to MRSA) were randomized to receive telavancin 10 mg/kg IV once daily. The maximum allowable treatment period was 14 days.
- Vancomycin: Patients with complicated Gram-positive skin and skin structure infections (primarily due to MRSA) were randomized to receive vancomycin 1 Gram every 12 hours. The maximum allowable treatment period was 14 days.
Period: Overall Study
Arm/Group | Telavancin | Vancomycin
Started | 429 | 433
Completed | 387 | 387
Not Completed | 42 | 46
Not completed — Adverse Event | 1 | 1
Not completed — Death | 4 | 5
Not completed — Lost to Follow-up | 26 | 23
Not completed — Withdrawal by Subject | 5 | 8
Not completed — Protocol Violation | 1 | 2
Not completed — Other | 2 | 3
Not completed — Never received study treatment | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Telavancin | Vancomycin | Total
Number analyzed (Participants) | 426 | 429 | 855
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 337 | 357 | 694
  >=65 years | 89 | 72 | 161
Age, Continuous [Mean (Standard Deviation); unit: years] | 49 (17.3) | 48 (16.1) | 48 (16.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 196 | 181 | 377
  Male | 230 | 248 | 478
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 114 | 97 | 211
  Not Hispanic or Latino | 312 | 332 | 644
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Patients could indicate more than one racial category.
  Participants
    American Indian or Alaska Native | 3 | 2 | 5
    Asian | 7 | 9 | 16
    Native Hawaiian or Other Pacific Islander | 3 | 9 | 12
    Black or African American | 59 | 52 | 111
    White | 349 | 353 | 702
    More than one race | 4 | 3 | 7
    Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 306 | 316 | 622
  South Africa | 11 | 12 | 23
  Australia | 18 | 15 | 33
  Belgium | 2 | 0 | 2
  Croatia | 49 | 51 | 100
  Israel | 15 | 12 | 27
  Malaysia | 5 | 4 | 9
  Russian Federation | 20 | 19 | 39
Diabetes Status [Number; unit: Participants]
  Diabetic | 94 | 98 | 192
  Not diabetic | 332 | 331 | 663

OUTCOME MEASURES:

1. Primary Outcome: Clinical Response
Description: The Clinical Response for each patient was determined by the investigator by assessing a patient's clinical signs and symptoms at the specified evaluation compared with the Baseline evaluation. Cure: resolution of signs and symptoms associated with the skin infection present at study admission such that no further antibiotic therapy was necessary; Not Cured: inadequate response to study therapy; Indeterminate: unable to determine outcome.
Time Frame: 7-14 days following end of antibiotic treatment
Population: Data for the all-treated (AT) population are presented. the AT and clinically evaluable (CE) populations were considered co-primary.
Measure: Number; unit: participants
Arm/Group | Telavancin | Vancomycin
Number analyzed (Participants) | 426 | 429
participants
  Cure | 323 | 321
  Not cured | 52 | 58
  Indeterminate | 23 | 16
  Missing | 28 | 34
Statistical Analysis 1: Comparison: Telavancin vs Vancomycin; Test type: Non-Inferiority or Equivalence — Non-inferiority margin of 10% was specified based on historical regulatory precedent; p-values were not calculated in deference to confidence intervals; Risk Difference (RD) = 1.0, 95% CI [-4.8 to 6.8] — Statistical analysis applies to "cure"

ADVERSE EVENTS:
Arm/Group | Telavancin | Vancomycin
Serious Adverse Events (participants affected / at risk) | 31/426 | 27/429
Other Adverse Events (participants affected / at risk) | 358/426 | 335/429
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Telavancin (N=426) | Vancomycin (N=429)
Renal Failure Acute (Renal and urinary disorders) | 1 | 0
Myocardial Infarction (Cardiac disorders) | 2 | 0
Blood creatinine increased (Investigations) | 0 | 2
Drug Hypersensitivity (Immune system disorders) | 1 | 1
Hypotension (Vascular disorders) | 1 | 1
Mental Status Changes (Psychiatric disorders) | 1 | 0
Renal Insufficiency (Renal and urinary disorders) | 1 | 0
Deep Vein Thrombosis (Vascular disorders) | 2 | 0
Osteomyelitis (Infections and infestations) | 1 | 0
Peripheral Occlusive Disease (Vascular disorders) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Renal Impairment (Renal and urinary disorders) | 2 | 0
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Angina Pectoris (Cardiac disorders) | 1 | 0
Ankle Fracture (Injury, poisoning and procedural complications) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 2
Bradycardia (Cardiac disorders) | 1 | 1
Calculus Bladder (Renal and urinary disorders) | 1 | 0
Cardio-Respiratory Arrest (Cardiac disorders) | 0 | 1
Cerebrovascular Accident (Nervous system disorders) | 1 | 0
Chest Discomfort (General disorders) | 1 | 0
Chronic Obstructive Airways Disease Exacerbated (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 1
Injection Site Cellulitis (General disorders) | 1 | 0
International Normalised Ratio Increased (Investigations) | 1 | 0
Myocardial Ischaemia (Cardiac disorders) | 1 | 0
Ovarian Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pulmonary Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Schizophrenia, Paranoid Type (Psychiatric disorders) | 1 | 0
Systemic Inflammatory Response Syndrome (General disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Urinary Tract Infection (Renal and urinary disorders) | 0 | 1
Varicose Vein Ruptured (Vascular disorders) | 1 | 0
Ventricular Arrhythmia (Cardiac disorders) | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 2
Bacteraemia (Infections and infestations) | 0 | 1
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Coma Hepatic (Nervous system disorders) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Non-Cardiac Chest Pain (General disorders) | 0 | 1
Ovarian Cyst (Reproductive system and breast disorders) | 0 | 1
Pelvic Infection (Infections and infestations) | 0 | 1
Post-Procedural Haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Procedural Hypotension (Injury, poisoning and procedural complications) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Renal Vessel Disorder (Renal and urinary disorders) | 0 | 1
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 1
White Blood Cell Count Increased (Blood and lymphatic system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Telavancin (N=426) | Vancomycin (N=429)
Anemia (Blood and lymphatic system disorders) | 12 | 8
Angina Pectoris (Cardiac disorders) | 5 | 1
Bradycardia (Cardiac disorders) | 2 | 5
Cardiac failure congestive (Cardiac disorders) | 5 | 2
Palpitations (Cardiac disorders) | 6 | 3
Vision blurred (Eye disorders) | 5 | 3
Abdominal Distension (Gastrointestinal disorders) | 5 | 4
Abdominal pain (Gastrointestinal disorders) | 11 | 17
Abdominal pain upper (Gastrointestinal disorders) | 5 | 8
Constipation (Gastrointestinal disorders) | 61 | 37
Diarrhoea (Gastrointestinal disorders) | 31 | 41
Dry Mouth (Gastrointestinal disorders) | 11 | 15
Dyspepsia (Gastrointestinal disorders) | 14 | 16
Loose stools (Gastrointestinal disorders) | 5 | 7
Nausea (Gastrointestinal disorders) | 128 | 95
Vomiting (Gastrointestinal disorders) | 78 | 50
Asthenia (General disorders) | 8 | 9
Fatigue (General disorders) | 19 | 21
Infusion site erythema (General disorders) | 7 | 9
Infusion site pain (General disorders) | 21 | 21
Infusion site phlebitis (General disorders) | 6 | 7
Infusion site pruritis (General disorders) | 5 | 9
Infusion site reaction (General disorders) | 7 | 7
Lethargy (General disorders) | 6 | 1
Non-Cardiac Chest Pain (General disorders) | 12 | 7
Oedema Peripheral (General disorders) | 8 | 11
Pain (General disorders) | 4 | 7
Pyrexia (General disorders) | 9 | 10
Rigors (General disorders) | 22 | 14
Fungal Infection (Infections and infestations) | 5 | 2
Osteomyelitis (Infections and infestations) | 5 | 4
Pneumonia (Infections and infestations) | 5 | 1
Urinary Tract Infection (Infections and infestations) | 6 | 4
Vaginal candidiasis (Infections and infestations) | 5 | 0
Vaginal mycosis (Infections and infestations) | 5 | 6
Anorexia (Metabolism and nutrition disorders) | 10 | 10
Decreased appetite (Metabolism and nutrition disorders) | 13 | 17
Hypoglycaemia (Metabolism and nutrition disorders) | 11 | 8
Hypokalemia (Metabolism and nutrition disorders) | 1 | 7
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 | 8
Back Pain (Musculoskeletal and connective tissue disorders) | 14 | 8
Muscle Cramp (Musculoskeletal and connective tissue disorders) | 5 | 6
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 8 | 7
Dizziness (Nervous system disorders) | 27 | 35
Dysgeusia (Nervous system disorders) | 156 | 31
Headache (Nervous system disorders) | 82 | 69
Hypoaesthesia (Nervous system disorders) | 3 | 5
Paresthesia (Nervous system disorders) | 3 | 5
Agitation (Psychiatric disorders) | 4 | 6
Anxiety (Psychiatric disorders) | 18 | 14
Confusional State (Psychiatric disorders) | 7 | 4
Insomnia (Psychiatric disorders) | 71 | 53
Restlessness (Psychiatric disorders) | 4 | 6
Dysuria (Renal and urinary disorders) | 7 | 5
Haematuria (Renal and urinary disorders) | 6 | 0
Renal Insufficiency (Renal and urinary disorders) | 5 | 1
Urinary Incontinence (Renal and urinary disorders) | 6 | 3
Urinary Abnormality (Renal and urinary disorders) | 69 | 8
Genital Pruritis Female (Reproductive system and breast disorders) | 8 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 12 | 13
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10 | 7
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 15 | 13
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 5
Dry Skin (Skin and subcutaneous tissue disorders) | 6 | 11
Erythema (Skin and subcutaneous tissue disorders) | 6 | 13
Exanthem (Skin and subcutaneous tissue disorders) | 7 | 4
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 10 | 9
Pruritis (Skin and subcutaneous tissue disorders) | 25 | 58
Pruritis generalized (Skin and subcutaneous tissue disorders) | 19 | 40
Rash (Skin and subcutaneous tissue disorders) | 17 | 23
Rash generalized (Skin and subcutaneous tissue disorders) | 1 | 9
Hot Flush (Vascular disorders) | 2 | 7
Hypertension (Vascular disorders) | 6 | 7
Hypotension (Vascular disorders) | 12 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less